CLINICAL TRIAL: NCT06496373
Title: Clinical Study of XP-004 Personlaized mRNA Vaccine Combined With PD-1 Inhibitor as Adjuvant Therapy for Postoperative Pancreatic Cancer
Brief Title: Clinical Study of mRNA Vaccine Combined With PD-1 Inhibitor as Adjuvant Therapy for Postoperative Pancreatic Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Shanghai Xinpu BioTechnology Company Limited (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023PCV004
Record Dates: First submitted 2024-06-18; First posted 2024-07-11 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Cancer Resectable; Chemotherapy-intolerant
Keywords: Personalized; Neoantigen; Pancreatic cancer; Postoperative adjuvant therapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoantigen based vaccines + PD-1 inhibitor (Experimental): A sequential treatment of single/fixed target mRNA vaccines (4 cycles) followed by Personalised mRNA vaccines (9 cycles), in combination with PD-1 inhibitor treatment every 3 weeks, 3 weeks as a treatment cycle, a total of 13 cycles.
  Interventions: Biological: Fixed neoantigen tumor vaccine; Biological: personalized neoantigen tumor vaccine; Drug: PD-1 inhibitor

INTERVENTIONS:
Biological: Fixed neoantigen tumor vaccine — Single/Fixed neoantigen mRNA vaccine includes pancreatic cancer driver mutations such as KRAS G12D, G12V, G12R, G12C, etc. Each vaccine has one neoantigen encoded by mRNA. Total of 4 cycles, 3 weeks each cycle.
Biological: personalized neoantigen tumor vaccine — personalized neoantigen tumor vaccine include 5-20 neoantigens selected based on WES/RNA-seq of patients' tumor sample during surgery. Total of 9 cycles after finishing the first 4 cycles of fixed neoantigen tumor vaccine.
Drug: PD-1 inhibitor — Toripalimab

SUMMARY:
This study primarily aims to assess the safety and tolerability of XP-004 personalized mRNA vaccines encoding tumor neoantigens combined with PD-1 inhibitor as adjuvant therapy for chemotherapy-intolerant patients following radical pancreatic cancer resection.

Secondary objectives focus on evaluating preliminary efficacy through three parameters: 1) XP-004-induced antigen-specific CD4+/CD8+ T cell activation levels, 2) recurrence-free survival (RFS), and 3) overall survival (OS) in post-operative pancreatic cancer patients receiving this combination therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily signed written informed consent files,Able to comply with the study protocol, in the investigator's judgment
2. Subjects must be >/= 18 years of age at time of informed consent, regardless of gender
3. Patients who have been confirmed by pathology to have pancreatic malignant tumors and have undergone radical surgery for pancreatic malignant tumors for 1-3 months
4. No copy number variations (CNVs) or loss of heterozygosity (Loss-of heterozygosity, LOH) were found in HLA-related genes and chromosomal regions by gene sequencing
5. Histologically confirmed pancreatic cancer samples underwent WES and RNA-seq analyses. Bioinformatics prediction identified at least one neoantigen effectively presented by the patient's HLA type, including those derived from KRAS or TP53 mutations.
6. According to the investigator's assessment, the patient is unable to tolerate chemotherapy, such as the score of the Eastern Cooperative Oncology Group (ECOG) Performance Scale ≥ 2 points

Exclusion Criteria:

1. Has had chemotherapy, traditional Chinese medicine with antitumor indications, or other antitumor therapies deemed to conflict with the current treatment by the investigator within 4 weeks prior to the first administration of the study drug
2. History of interstitial lung disease (ILD), pulmonary fibrosis
3. Other serious and/or uncontrollable diseases, which may affect the subject's participation in this study, include but not limited to a) a history of severe drug allergy, or is known to be allergic to any tumor vaccine and PD-1 inhibitor formulation components or has had severe allergic reactions to other monoclonal antibodies in the past, b) A history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases
4. Researchers believe that there are other reasons that are not suitable for participating in clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Drug related toxicity | 18 months
  Percentage Participants with Adverse Events (AEs) by severity According to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0

SECONDARY OUTCOMES:
Recurrence-free survival (RFS) | Up to 18 months
  Recurrence-free survival of Personalized mRNA Tumor Vaccine
overall survival (OS) | Up to 18 months
  Overall Survival of Personalized mRNA Tumor Vaccine
Reaction of antigen-specific T cells in peripheral blood | Up to 18 months
  personalized tumor vaccine induced neoantigen-specific CD4+ and CD8+ T lymphocyte responses

CONTACTS AND LOCATIONS:
Overall Officials: Baiyong Shen, M.D&Ph.D, Study Director — Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No